CLINICAL TRIAL: NCT03997331
Title: A Phase 1, Randomized Controlled Trial of the Chronicare Disease Management Program in Subjects With Type 2 Diabetes (Chronicare-T2D)
Brief Title: Chronicare for Type 2 Diabetes (Chronicare-T2D)
Acronym: CRX-T2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: QuiO (Industry)
Collaborators: SHL Medical (Unknown); MidMichigan Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1433742-2
Record Dates: First submitted 2019-06-20; First posted 2019-06-25 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects in the Intervention arm will receive the following:
  1. Automated in-app messages containing behavioral and educational content that is tailored to each subject based on an assessment of their entry survey results and on their adherence and glucose data. (Behavioral Support Engine).
  2. Targeted in-app messages and phone calls from clinicians or as designated by the Investigator (through the CRx Care app) based on the subject's adherence and glucose data.
  3. Push notifications that alert the subject that it is time to complete a regimen event (ie take medication or take a fasting blood glucose reading).
  4. Push notifications that alert the subject that they have missed a scheduled regimen event.
  5. In-app messages containing adjustments to the subject's insulin glargine dose when the Investigator(s) approves an adjustment in the CRx Care App. (Treatment Support Engine).
  Interventions: Other: CRx Health; Other: Chronicare
- Control (Active Comparator): Subjects in the Control arm will receive the CRx Health solution for self-management of chronic conditions.
  Interventions: Other: CRx Health

INTERVENTIONS:
Other: CRx Health — CRx Health is a connected health solution comprised of connected devices (InsulCheck, a Bluetooth-enabled pill bottle cap, and a Bluetooth-enabled glucometer) paired to a mobile smartphone app (CRx Health).
Other: Chronicare — Chronicare is a disease management program comprising self-management data from the CRx Health solution syncing to an automated support system (Intervention Engine) and a remote care application (CRx Care) used by a team of clinicians to remotely monitor and support patients.
  Arms: Intervention

SUMMARY:
This single-blind, single-center, randomized, controlled trial is designed to evaluate the utility of the Chronicare Disease Management Program in the management of subjects with T2D who are being treated with insulin glargine and metformin. The Chronicare Solution comprises connected devices (a Bluetooth-enabled insulin pen sensor, a Bluetooth-enabled medication container, and a Bluetooth-enabled glucometer), a mobile smartphone app (CRx Health), an automated support system (Intervention Engine), and a remote care application (CRx Care) used by a team of clinicians to monitor and support patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 75 years of age, inclusive, at Screening.
* Diagnosed with T2D
* Have a baseline HbA1c level between 7.5% and 10.0%, inclusive, while receiving insulin glargine and metformin.
* Prescribed insulin glargine and an oral diabetes medication for ≥ 6 months prior to Screening.
* The ability to follow an evening dosing schedule for insulin glargine.
* Have an eGFR level >30 L/min, inclusive, according to their most recent measurement.
* If female, must be post-menopausal or surgically sterile, or be established on (≥ 3 months prior to Screening) and agree to continue to use the same highly effective method of birth control throughout the study. Females must agree to avoid pregnancy during their participation in the study.
* Able to comprehend and give informed consent.
* Able to comply with the requirements of the study, which include being able to speak and read English, and to complete the full sequence of protocol-related procedures.

Exclusion Criteria:

* Females who are pregnant (positive pregnancy test at Screening), lactating, or if having reproductive potential, are considered potentially unreliable with respect to contraceptive practice.
* Have type 1 diabetes.
* Have had or have a malignant neoplasm within the past five years.
* Undergoing chronic or recurrent treatment with systemic corticosteroids or niacin treatment for hyperlipidemia.
* Use of one or more of the following agents affecting glycemic control:

mifepristone, GLP-1RA, or any insulin other than insulin glargine.

* Concurrent treatment with experimental drugs or participation in another clinical trial with any investigational drug within 30 days or 5 half-lives, whichever is greater, prior to study start.
* Unable or unwilling to follow the evening insulin glargine regimen required by the titration protocol (once daily dose must be scheduled between 5pm and 12am).
* Blood transfusions or severe blood loss in the last 3 months.
* Any other unspecified reason that, in the opinion of the Investigator (or designee) or Sponsor, makes the subject unsuitable for enrollment.
* Active diagnosis of hypoglycemic unawareness.
* Hypoglycemia (blood glucose <70 mg/dl with or without symptoms) greater than one episode per week (on average)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Day 0 - Day 120
  The primary endpoint is the difference in the reduction in HbA1c for each subject by treatment group (Intervention vs. Control), assessed by the mean reduction across all subjects in each treatment group.

SECONDARY OUTCOMES:
Fasting Blood Glucose | Day 0 - Day 120
  Fasting blood glucose level (Intervention vs. Control), measured by the proportion of measurements of self-reported fasting blood glucose within the range of 70-110 mg/dL for subjects in each study arm
Mean Duration of Time to Reach Optimal Insulin Glargine Dose | Up to 120 days
  Optimal insulin glargine dose (Intervention vs. Control), measured by the mean duration of time elapsed prior to reaching a mean self-reported fasting blood glucose value of 70-110 mg/dL over a 7-day period.
Proportion of Patients Reaching Optimal Insulin Glargine Dose | Day 120
  Optimal insulin glargine dose (Intervention vs. Control), measured by the proportion of patients reaching a mean self-reported fasting blood glucose value of 70-110 mg/dL over a 7-day period.
Median Adherence to Insulin Glargine | Day 0 - Day 120
  Insulin glargine adherence by treatment group (Intervention vs. Control), assessed by median adherence computed as percentage of doses taken on time (±2h dosing window).
Median Adherence to Metformin | Day 0 - Day 120
  Metformin adherence by treatment group (Intervention vs. Control), assessed by median adherence computed as percentage of doses taken on time (±2h dosing window).

CONTACTS AND LOCATIONS:
Overall Officials: Sujay Madduri, MD, Principal Investigator — MidMichigan Health; Alexander Dahmani, Study Chair — QuiO Technologies
Locations (1):
- Clinical Research Department, Midland, Michigan, United States